CLINICAL TRIAL: NCT03929562
Title: Alcohol Screening and Pre-Operative Intervention Research Study
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anne Fernandez, Assistant Professor of Psychiatry, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HUM00156743; 5K23AA023869 (NIH)
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Drinking
Keywords: Elective Surgery
MeSH Terms: conditions — Alcohol Drinking | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief advice (Active Comparator): One brief advice session, resource brochure, standard of care, and an infographic about alcohol and surgical health at patient's pre-existing pre-operative clinical visit.
  Interventions: Behavioral: Brief advice
- Health coaching (Experimental): Two health coaching sessions, resource brochure, standard of care
  Interventions: Behavioral: Health coaching

INTERVENTIONS:
Behavioral: Brief advice — One 10-minute brief advice session
  Arms: Brief advice
Behavioral: Health coaching — Two 45-minute health coaching sessions will use a non-confrontation motivational interviewing (MI) style. Intervention delivery will include expressing concern about unhealthy drinking, providing feedback linking alcohol use and health (related to surgery and general health), advising the patient regarding abstinence or alcohol use reduction, and working with the patient to set a drinking goal if he/she is ready to change. We will also include a personalized feedback component to address the links between pre-operative alcohol use and postoperative morbidity/mortality.
  Arms: Health coaching

SUMMARY:
This study aims to learn more about how to improve patients' health before and after a scheduled surgery by examining acceptability and initial efficacy of pre-operative alcohol use reduction interventions.

DETAILED DESCRIPTION:
The study is a randomized clinical pilot trial that assesses preliminary intervention efficacy of a two-session health coaching intervention relative to brief advice among pre-operative elective surgical patients and evaluates intervention acceptability. Study subjects will be outpatients at a large health system in the midwestern United States and fulfill the study's inclusion criteria. Subjects will be randomized to one of two intervention conditions: Health Coaching or Brief Advice.

ELIGIBILITY:
Inclusion Criteria:

* Referred for elective or semi-elective surgery or pre-operative assessment in the next 120 days
* Meet criteria for "risky drinking" as defined by study staff

Exclusion Criteria:

* Displays or shows evidence of psychotic symptoms
* Undergoing surgeries that commonly require local anesthesia only

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fernandez, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers will plan to share individual participant data that underlies the results reported in an article, after deidentification (text, tables, figures, and appendices), Study protocol, and Informed Consent Form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Chapman L, Ren T, Solka J, Bazzi AR, Borsari B, Mello MJ, Fernandez AC. Reducing Alcohol Use Before and After Surgery: Qualitative Study of Two Treatment Approaches. JMIR Perioper Med. 2023 Jul 26;6:e42532. doi: 10.2196/42532. PMID 37494103

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 of 65 enrolled participants were not assigned to groups because they did not meet eligibility requirements after enrollment (i.e. surgery cancelation).
Groups:
- Brief Advice: One 10-minute educational and feedback intervention delivered 4 weeks prior to surgery.
- Health Coaching: Two 45-minute Health Coaching sessions delivered 4 weeks and 2 weeks prior to surgery, respectively. The sessions were based on the principles of collaborative care, motivational interviewing, and the Health Belief Model. Intervention delivery included education about alcohol use and surgical risk, providing feedback linking alcohol use and health (related to surgery and general health), advising the patient regarding abstinence or alcohol use reduction, and working with the patient to set a drinking goal if he/she was ready to change.
Period: From Baseline to 1 Month Follow Up
Arm/Group | Brief Advice | Health Coaching
Started | 26 | 25
Completed | 22 | 24
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Period: 1 Month Follow Up to 4 Month Follow Up
Arm/Group | Brief Advice | Health Coaching
Started | 22 | 24
Completed | 20 | 24
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Advice | Health Coaching | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (13.9) | 49.4 (14.4) | 47.7 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Ethnicity | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 20 | 44
  Black | 0 | 2 | 2
  Asian | 1 | 1 | 2
  American Indian/Alaska Native | 0 | 1 | 1
  Other Race | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 25 | 51
Marital Status [Count of Participants; unit: Participants]
  Married | 16 | 12 | 28
  Not Married | 10 | 13 | 23
Highest Education [Count of Participants; unit: Participants]
  Some high school | 0 | 1 | 1
  High school/GED | 3 | 2 | 5
  Some college | 4 | 6 | 10
  College graduate | 15 | 11 | 26
  Post college | 4 | 5 | 9
Surgical Stay [Count of Participants; unit: Participants]
  Inpatient | 4 | 6 | 10
  Outpatient | 22 | 19 | 41
Surgical Service [Count of Participants; unit: Participants]
  Plastic | 11 | 12 | 23
  Orthopedic | 6 | 7 | 13
  Minimally Invasive | 5 | 2 | 7
  Endocrine | 1 | 1 | 2
  Gynecology | 1 | 1 | 2
  Urology | 1 | 1 | 2
  Colorectal | 1 | 0 | 1
  Hepatobiliary | 0 | 1 | 1
Alcohol Use Disorders Identification Test (AUDIT-C) Score [Mean (Standard Deviation); unit: units on a scale] — The three-item AUDIT-C assessed alcohol quantity, frequency, and heavy drinking days. The overall score ranges from 0 to 12, with zero reflecting no alcohol use and higher scores reflecting higher levels of alcohol use.
  units on a scale | 6.4 (1.4) | 6.2 (1.5) | 6.3 (1.5)
Drinks consumed per week [Mean (Standard Deviation); unit: Drinks consumed/week] | 13.8 (12.5) | 10.7 (7.8) | 12.3 (10.5)
Percentage of Days Abstinent [Mean (Standard Deviation); unit: Percentage] | 47.8 (33.8) | 52.8 (32.8) | 50.3 (33.0)
Percentage of Weeks Exceeding Moderate Drinking [Mean (Standard Deviation); unit: Percentage] | 54.1 (39.6) | 43.7 (38.9) | 49.0 (39.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Alcohol Weekly Use
Description: Average (i.e. mean) weekly alcohol use was assessed using the timeline followback measure. The timeline followback assesses alcohol use using a calendar format on which participants report the number of standard drinks they consumed each day during the assessment period. In the United States, one standard drink (or one alcoholic drink equivalent), is defined as any beverage containing 0.6 oz or 14 grams of pure alcohol.
Time Frame: Baseline through 4 months
Measure: Mean (Standard Deviation); unit: Drinks consumed/week
Arm/Group | Brief Advice | Health Coaching
Number analyzed (Participants) | 26 | 25
Drinks consumed/week
  1-Month Follow Up | 7.01 (3.12) | 6.07 (2.13)
  4-Month Follow Up | 8.15 (3.08) | 6.44 (1.91)

2. Secondary Outcome: Acceptability of Intervention as Measured by the Post-intervention Evaluation.
Description: Interventions will be considered 'acceptable' if the average acceptability rating reaches a threshold of 3 or more on a 4-point Likert scale where a score of 4 is most acceptable.
  Satisfaction
  1. Quite dissatisfied
  2. Mildly dissatisfied
  3. Mostly satisfied
  4. Very satisfied
Time Frame: Weeks 1-6, Immediately following intervention
Population: Among the Brief Advice participants only 23 completed this survey.
Measure: Count of Participants; unit: Participants
Groups:
- Health Coaching Session 1: This 45-minute Health Coaching session was delivered 4 weeks prior to surgery. The session was based on the principles of collaborative care, motivational interviewing, and the Health Belief Model. Session 1 focused on alcohol use and surgical risk reduction in the 4 weeks prior to surgery. Intervention delivery included education about alcohol use and surgical risk, providing feedback linking alcohol use and health (related to surgery and general health), advising the patient regarding abstinence or alcohol use reduction, and working with the patient to set a drinking goal if he/she was ready to change.
- Health Coaching Session 2: This 45-minute Health Coaching session was delivered 2 weeks prior to surgery. The session was based on the principles of collaborative care, motivational interviewing, and the Health Belief Model. Session 2 focused on alcohol use and surgical risk reduction in the 6 weeks after surgery. Intervention delivery included education about alcohol use and surgical risk, reviewing change since session 1, providing feedback linking alcohol use and health (related to surgery and general health), advising the patient regarding abstinence or alcohol use reduction, and working with the patient to set or maintain a drinking goal if he/she was ready to change.
Arm/Group | Brief Advice | Health Coaching Session 1 | Health Coaching Session 2
Number analyzed (Participants) | 23 | 24 | 24
Participants
  Mostly Satisfied (3) | 8 | 4 | 1
  Very Satisfied (4) | 15 | 20 | 23

ADVERSE EVENTS:
Time Frame: 4 Months
Arm/Group | Brief Advice | Health Coaching
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/26 | 3/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief Advice (N=26) | Health Coaching (N=25)
Post-op Surgical complications, Surgical and Medical Procedures (Injury, poisoning and procedural complications) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT03929562/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03929562/ICF_001.pdf